CLINICAL TRIAL: NCT03921645
Title: Use of Aaerosol Combined With Intravenous Antibiotics for the Treatment of Multidrug Resistant GNB Pneumonia
Acronym: ACAMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Sheng Wang MD PhD, Director, Principal investigator, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ACAMP
Record Dates: First submitted 2017-11-20; First posted 2019-04-19 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Ventilator Associated Pneumonia; Multi-antibiotic Resistance
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- aerosol combined group (Experimental): aerosol combined intravenous antibiotics group，amikacin 15mg/kg, qd
  Interventions: Drug: aerosol antibiotics
- No intervention group (No Intervention): this group follow the usual treatment without any intervention

INTERVENTIONS:
Drug: aerosol antibiotics — use of inhaled Antibacterial drug combined with intravenous antibiotics to treatment multiple drug resistance GNB ventilator associated pneumonia.
  Arms: aerosol combined group

SUMMARY:
To investigate use of aerosol combined with intravenous antibiotics for the treat of multi-drug resistance gram negative bacterias diagnosed ventilator-associated pneumonia in intensive care unit in a hospital.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) refers to the endotracheal tube or tracheostomy patients pneumonia after 48h of mechanical ventilation, mechanical ventilation is one of the most common and most serious complications, hospital acquired is An important cause of pneumonia. According to the onset time of VAP, VAP can be divided into early-onset VAP and late-onset VAP. The time limit is mechanical ventilation for 4 days, in which early-onset VAP (mechanical ventilation ≤ 4d) is mainly caused by pathogens sensitive to most antibacterial drugs (such as methicillin-sensitive Staphylococcus aureus, Streptococcus pneumoniae, etc.); late-onset VAP ≥ 5D occur during mechanical ventilation, mainly caused by multi-drug resistant (multi-drug resistance, MDR) (such as P. aeruginosa, Acinetobacter baumannii, methicillin-resistant Staphylococcus aureus). Some early-onset VAPs can also be caused by MDR. Therefore, MDR has become the main pathogen of VAP, especially Gram-negative bacilli. Studies have shown that VDR caused by MDR has a mortality rate of 76% and an attributable mortality rate of 20-30%. Such bacteria are not sensitive to commonly used antibacterial drugs in the clinic, and sensitive antibiotics, such as aminoglycosides, have a large systemic side effect, thereby limiting clinical use. Therefore, in theory, nebulized inhaled sensitive antibiotics can achieve high drug concentrations in lung tissue, and lower blood concentrations can avoid or reduce systemic side effects.

ELIGIBILITY:
Inclusion Criteria:

・After 48 hours of mechanical ventilation diagnosed VAP.

Exclusion Criteria:

* Maternal
* who not meet the age limits,
* used amikacin within 15 days,
* allergic to amikacin,
* APACHE II score > 35,
* severe neutropenia unrelated to sepsis or meningitis,
* unable to retain specimens

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
CPIS score changes | 14 days
  use clinical pulmonary infection score scale to evaluate score change from baseline for every patient
renal function changes | 14 days
  record changes in renal function assessed by SCr, blood urea nitrogen,etc.

SECONDARY OUTCOMES:
ventilator free days in 14 days | 14 days
  record number of days with no ventilator support from day 1 through day 14
14-day mortality rate | 14 days
  rate of mortality from day 1 to day 14
Drug resistance induction rate | 14 days
  Drug resistance induction rate is The number of cases of antibiotic-resistant species from the previous increase divided by the total number of patients included

CONTACTS AND LOCATIONS:
Overall Officials: hao liu, master, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai tenth people's hospital, Shanghai, Shanghai Municipality, China